CLINICAL TRIAL: NCT01362491
Title: Ibuprofen Sodium Tension Headache Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-11-16; B3411007
Record Dates: First submitted 2011-05-19; First posted 2011-05-30 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Pain
Keywords: Headache
MeSH Terms: conditions — Pain; Headache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Ibuprofen Sodium
- Treatment B (Active Comparator)
  Interventions: Drug: Standard Ibuprofen
- Treatment C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen Sodium — Single-dose of ibuprofen sodium tablets (equal to 400 mg ibuprofen)
  Arms: Treatment A
Drug: Standard Ibuprofen — Single-dose of standard ibuprofen tablets (400mg)
  Arms: Treatment B
Drug: Placebo — Single-dose of placebo
  Arms: Treatment C

SUMMARY:
This study will compare the ability of a single-dose of a novel ibuprofen formulation to relieve pain compared to placebo and standard ibuprofen in the treatment of tension-type headache

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years to 65 years of age
* A diagnosis of an episodic tension-type headache, as defined by the International Headache Society

Exclusion Criteria:

* Pregnancy or breast-feeding
* Alcohol or substance abuse
* Any serious medical or psychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Packman E, Leyva R, Kellstein D. Onset of analgesia with ibuprofen sodium in tension-type headache: a randomized trial. J Pharm Health Care Sci. 2015 Apr 2;1:13. doi: 10.1186/s40780-015-0012-9. eCollection 2015. PMID 26819724
- [Derived] Jayawardena S, Leyva R, Kellstein D. Safety of a novel formulation of ibuprofen sodium compared with standard ibuprofen and placebo. Postgrad Med. 2015 Jan;127(1):33-7. doi: 10.1080/00325481.2015.993268. Epub 2014 Dec 15. PMID 25526232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AH-11-16&StudyName=Ibuprofen%20Sodium%20Tension%20Headache%20Study%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen Sodium: Single oral dose of 2 ibuprofen sodium 256 mg tablets, equivalent to 400 mg ibuprofen along with single oral dose of 2 placebo tablets matched to ibuprofen (Motrin IB) 200 mg tablet.
- Ibuprofen (Motrin IB): Single oral dose of 2 ibuprofen (Motrin IB) 200 mg tablets (total dose to 400 mg ibuprofen) along with single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 mg tablet.
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen [Motrin ibuprofen (IB)] 200 milligram (mg) tablet along with single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 mg tablet.
Period: Overall Study
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Started | 91 | 89 | 46
Completed | 90 | 89 | 46
Not Completed | 1 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo | Total
Number analyzed (Participants) | 91 | 89 | 46 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (14.3) | 44.8 (13.5) | 39.9 (15.2) | 42.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 30 | 149
  Male | 31 | 30 | 16 | 77
Pain Severity Score [Number; unit: participants] — Pain severity score was assessed on a 4-point categorical scale. Total possible pain severity was 0 to 3, where 0 = none, 1 = mild, 2 = moderately severe and 3 = severe.
  participants
    Moderately Severe | 73 | 70 | 36 | 179
    Severe | 18 | 19 | 10 | 47

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference From 0-3 Hours (SPRID 0-3) for Ibuprofen Sodium Versus Placebo Tablet
Description: SPRID:time-weighted sum of pain relief rating combined with pain intensity difference (PRID) over 3 hours. SPRID score range:-3 (worst) to 21 (best) for SPRID 0-3. PRID: sum of pain intensity differences (PID) and pain relief rating(PRR) at each time point. PRID score range: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3 (best). PRR:assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0-3 Hours
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Placebo
Number analyzed (Participants) | 91 | 46
units on scale | 9.6 (4.8) | 3.5 (4.2)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; Treatment difference (Ibuprofen sodium-placebo) and 95 percent (%) confidence interval (CI): based on LS means from analysis of variance (ANOVA). Type I error was controlled at 0.05 significance level (2-sided) by declaring pair wise comparisons significant only if overall treatment effect among 3 treatment groups was significant and testing in a sequential order Ibuprofen sodium versus (vs.) placebo for SPRID 0-3 then Ibuprofen sodium vs. Ibuprofen (Motrin IB) for time to meaningful relief; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline Pain Severity Rating (PSR) and gender terms; Least-Square (LS) mean difference = 6.11, 95% CI 2-sided [4.49 to 7.73]

2. Primary Outcome: Time to Onset of Meaningful Relief for Ibuprofen Sodium Versus Ibuprofen (Motrin IB) Tablet
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment the participant first began to experience meaningful relief. It was also considered achieved if the participant stated "meaningful relief" at the time the first stopwatch was depressed. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 91 | 89
minutes | 40.6 [36.7 to 46.8] | 48.5 [45.5 to 53.5]
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); Hazard Ratio (HR) and corresponding 95% CI were calculated based on the Wald statistic from the proportional hazards (PH) model. Type I error was controlled at 0.05 significance level (2-sided) by declaring pair wise comparisons significant only if overall treatment effect among 3 treatment groups was significant and testing in a sequential order Ibuprofen sodium vs. placebo for SPRID 0-3 then Ibuprofen sodium vs. Ibuprofen (Motrin IB) for time to meaningful relief; Test type: Superiority or Other; p = 0.253, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline Pain Severity Rating (PSR) and gender terms; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.88 to 1.65]

3. Secondary Outcome: Time to Onset of Meaningful Relief: Remaining Comparisons
Description: as for outcome 2
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
minutes | 40.6 [36.7 to 46.8] | 48.5 [45.5 to 53.5] | NA [NA to NA] — Data was not summarized as the median time to onset of meaningful relief was >180 minutes (>3 hours) for placebo group and therefore the 95% CI was not estimable.
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline Pain Severity Rating (PSR) and gender terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 4.38, 95% CI 2-sided [2.69 to 7.14]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 3.64, 95% CI 2-sided [2.23 to 5.94]

4. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment the participant first began to experience any relief. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered. First perceptible relief was considered confirmed by meaningful relief if the participant achieved both "first perceptible" and "meaningful" relief by either depressing the second stopwatch or by indicating that his/her "first perceptible" relief was also "meaningful".
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
minutes | 36.9 [34.5 to 40.7] | 43.6 [40.1 to 48.4] | NA [NA to NA] — Data was not summarized as the median time to first perceptible relief confirmed by meaningful relief was >180 minutes (>3 hours) for placebo group and therefore the 95% CI was not estimable.
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 4.68, 95% CI 2-sided [2.87 to 7.64]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 3.88, 95% CI 2-sided [2.38 to 6.34]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.247, Proportional hazards model — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.88 to 1.66]

5. Secondary Outcome: Pain Relief Rating (PRR)
Description: PRR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: 1, 2 & 3 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  1 hour | 1.5 (1.0) | 1.6 (1.0) | 0.3 (0.7)
  2 hours | 2.3 (1.0) | 2.2 (1.0) | 1.0 (1.0)
  3 hours | 2.8 (1.3) | 2.9 (1.2) | 1.2 (1.2)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline Pain Severity Rating (PSR) and gender terms. Statistical testing was done at 5% significance level (2-sided); Least Square (LS) mean difference = 1.26, 95% CI 2-sided [0.92 to 1.59]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; 1 hour: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.27, 95% CI 2-sided [0.93 to 1.61]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.943, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.01, 95% CI 2-sided [-0.29 to 0.27]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.25, 95% CI 2-sided [0.89 to 1.62]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; 2 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.22, 95% CI 2-sided [0.85 to 1.59]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.847, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.03, 95% CI 2-sided [-0.27 to 0.33]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Placebo; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.59, 95% CI 2-sided [1.14 to 2.05]
Statistical Analysis 8: Comparison: Ibuprofen (Motrin IB) vs Placebo; 3 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.68, 95% CI 2-sided [1.22 to 2.13]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - (Ibuprofen IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.663, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.08, 95% CI 2-sided [-0.46 to 0.29]

6. Secondary Outcome: Pain Intensity Difference (PID)
Description: PID was derived by subtracting the pain severity score at a given post-dosing time point [pain severity score range 0 (none) to 3 (severe)] from the baseline score [Baseline pain severity score range 2 (moderately severe) to 3 (severe)]. Total possible score range for PID: -1 (worst) to 3 (best).
Time Frame: 1, 2 & 3 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  1 hour | 0.7 (0.5) | 0.7 (0.6) | 0.2 (0.4)
  2 hours | 1.0 (0.6) | 1.0 (0.5) | 0.4 (0.6)
  3 hours | 1.3 (0.9) | 1.4 (0.8) | 0.5 (0.8)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.54, 95% CI 2-sided [0.37 to 0.72]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.51, 95% CI 2-sided [0.33 to 0.69]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.651, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.03, 95% CI 2-sided [-0.11 to 0.18]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.62, 95% CI 2-sided [0.42 to 0.81]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.65, 95% CI 2-sided [0.46 to 0.85]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.669, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.03, 95% CI 2-sided [-0.19 to 0.13]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.84, 95% CI 2-sided [0.57 to 1.11]
Statistical Analysis 8: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.94, 95% CI 2-sided [0.67 to 1.21]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.396, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.10, 95% CI 2-sided [-0.32 to 0.13]

7. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference (PRID)
Description: PRID was sum of PID and PRR at each post-dosing time point. The overall possible score range, for PRID was -1 (worst) to 7 (best). PID was derived by subtracting the pain severity score at a given post-dosing time point [pain severity score range 0 (none) to 3 (severe)] from the baseline score [Baseline pain severity score range 2 (moderately severe) to 3 (severe)]. Total possible score range for PID: -1 (worst) to 3 (best). PRR was assessed on 5-point categorical pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 1, 2 & 3 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  1 hour | 2.3 (1.4) | 2.2 (1.6) | 0.5 (1.0)
  2 hours | 3.2 (1.6) | 3.2 (1.5) | 1.4 (1.5)
  3 hours | 4.1 (2.1) | 4.3 (2.0) | 1.7 (1.9)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.80, 95% CI 2-sided [1.30 to 2.30]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.78, 95% CI 2-sided [1.28 to 2.28]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.911, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.02, 95% CI 2-sided [-0.39 to 0.43]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.87, 95% CI 2-sided [1.33 to 2.41]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.88, 95% CI 2-sided [1.34 to 2.42]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.982, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.00, 95% CI 2-sided [-0.45 to 0.44]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.44, 95% CI 2-sided [1.72 to 3.15]
Statistical Analysis 8: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.61, 95% CI 2-sided [1.90 to 3.33]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 6, analysis 9]; Test type: Superiority or Other; p = 0.547, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.18, 95% CI 2-sided [-0.77 to 0.41]

8. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID)
Description: SPID: time-weighted sum of PID over 2 and 3 hours. SPID score range was -2(worst) to 6 (best) for SPID 0-2 and -3 (worst) to 9 (best) for SPID 0-3. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3 (best).
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  SPID 0-2 | 1.7 (1.0) | 1.7 (1.0) | 0.5 (0.9)
  SPID 0-3 | 3.0 (1.8) | 3.1 (1.6) | 1.0 (1.6)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; SPID 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.16, 95% CI 2-sided [0.83 to 1.50]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; SPID 0-2: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 1.17, 95% CI 2-sided [0.83 to 1.50]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPID 0-2: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.992, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.00, 95% CI 2-sided [-0.28 to 0.27]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; SPID 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.01, 95% CI 2-sided [1.43 to 2.58]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; SPID 0-3: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.10, 95% CI 2-sided [1.53 to 2.68]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPID 0-3: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.684, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.10, 95% CI 2-sided [-0.57 to 0.38]

9. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR)
Description: TOTPAR: time-weighted sum of PRR over 2 and 3 hours. TOTPAR score range was 0 (worst) to 8 (best) for TOTPAR 0-2 and 0 (worst) to 12 (best) for TOTPAR 0-3. PRR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  TOTPAR 0-2 | 3.8 (1.9) | 3.8 (1.9) | 1.3 (1.5)
  TOTPAR 0-3 | 6.6 (3.1) | 6.6 (3.0) | 2.5 (2.7)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; TOTPAR 0-2: Treatment difference (Ibuprofen Sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.51, 95% CI 2-sided [1.85 to 3.17]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; TOTPAR 0-2: Treatment difference [Ibuprofen (Motrin IB) - Placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 2.49, 95% CI 2-sided [1.83 to 3.15]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); TOTPAR 0-2: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.943, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.02, 95% CI 2-sided [-0.52 to 0.56]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; TOTPAR 0-3: Treatment difference (Ibuprofen Sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 4.10, 95% CI 2-sided [3.03 to 5.18]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; TOTPAR 0-3: Treatment difference [Ibuprofen (Motrin IB) - Placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 4.17, 95% CI 2-sided [3.09 to 5.24]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); TOTPAR 0-3: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.888, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.06, 95% CI 2-sided [-0.95 to 0.82]

10. Secondary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference (SPRID)
Description: SPRID: time-weighted sum of PRID over 2 and 3 hours. SPRID score range was -2(worst) to 14(best) for SPRID 0-2 and -3 (worst) to 21 (best) for SPRID 0-3. PRID: sum of PID and PRR at each time point. Total score range for PRID: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3(best), PRR: assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
units on scale
  SPRID 0-2 | 5.5 (2.8) | 5.5 (2.8) | 1.8 (2.4)
  SPRID 0-3 | 9.6 (4.8) | 9.8 (4.6) | 3.5 (4.2)
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; SPRID 0-2: Treatment difference (Ibuprofen Sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 3.67, 95% CI 2-sided [2.71 to 4.64]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; SPRID 0-2: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 3.66, 95% CI 2-sided [2.68 to 4.63]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPRID 0-2: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.964, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 0.02, 95% CI 2-sided [-0.78 to 0.82]
Statistical Analysis 4: Comparison: Ibuprofen (Motrin IB) vs Placebo; SPRID 0-3: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = 6.27, 95% CI 2-sided [4.65 to 7.89]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPRID 0-3: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.812, ANOVA — [p-value comment as in outcome 5, analysis 1]; Least Square (LS) mean difference = -0.16, 95% CI 2-sided [-1.49 to 1.17]

11. Secondary Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief evaluated by stopping a second stopwatch labeled 'meaningful relief' at the moment the participant first began to experience meaningful relief. It was also considered achieved if the participant stated "meaningful relief" at the time the first stopwatch was depressed. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0.5, 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
percentage of participants
  0.5 hours | 12.1 | 4.5 | 0
  1 hour | 71.4 | 65.2 | 13
  2 hours | 85.7 | 86.5 | 39.1
  3 hours | 85.7 | 86.5 | 45.7
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel — p-value was calculated using CMH test which was adjusted for baseline Pain Severity Rating (PSR) and gender. Statistical testing was done at 5% significance level (2-sided); Difference in proportion = 12.02, 95% CI 2-sided [5.27 to 18.77]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; 0.5 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.146, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 4.50, 95% CI 2-sided [0.13 to 8.88]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 0.5 hours: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.064, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 7.62, 95% CI 2-sided [-0.38 to 15.63]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 58.58, 95% CI 2-sided [44.96 to 72.21]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; 1 hour: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 52.31, 95% CI 2-sided [38.20 to 66.41]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.357, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 6.40, 95% CI 2-sided [-7.27 to 20.07]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Placebo; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 46.68, 95% CI 2-sided [30.43 to 62.93]
Statistical Analysis 8: Comparison: Ibuprofen (Motrin IB) vs Placebo; 2 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 47.59, 95% CI 2-sided [31.35 to 63.83]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.889, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.72, 95% CI 2-sided [-10.89 to 9.45]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Placebo; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 40.26, 95% CI 2-sided [23.85 to 56.68]
Statistical Analysis 11: Comparison: Ibuprofen (Motrin IB) vs Placebo; 3 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 41.19, 95% CI 2-sided [24.78 to 57.59]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen Sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.889, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.72, 95% CI 2-sided [-10.89 to 9.45]

12. Secondary Outcome: Cumulative Percentage of Participants With First Perceptible Relief
Description: Percentage of participants with first perceptible relief evaluated by stopping a stopwatch labeled 'first perceptible relief' at the moment the participant first began to experience any relief. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered. First perceptible relief was considered confirmed by meaningful relief if the participant achieved both "first perceptible" and "meaningful" relief by either depressing the second stopwatch or by indicating that his/her "first perceptible" relief was also "meaningful".
Time Frame: 0.5, 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
percentage of participants
  0.5 hours | 18.7 | 7.9 | 0
  1 hour | 76.9 | 74.2 | 15.2
  2 hours | 85.7 | 86.5 | 45.7
  3 hours | 85.7 | 86.5 | 45.7
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 18.58, 95% CI 2-sided [10.43 to 26.73]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.055, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 7.80, 95% CI 2-sided [2.14 to 13.46]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.033, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 10.91, 95% CI 2-sided [0.98 to 20.83]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 62.03, 95% CI 2-sided [48.65 to 75.41]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 59.44, 95% CI 2-sided [45.69 to 73.19]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.642, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 2.96, 95% CI 2-sided [-9.52 to 15.44]
Statistical Analysis 7: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 40.26, 95% CI 2-sided [23.85 to 56.68]
Statistical Analysis 8: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 8]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 41.19, 95% CI 2-sided [24.78 to 57.59]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; p = 0.889, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.72, 95% CI 2-sided [-10.89 to 9.45]
Statistical Analysis 10: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 40.26, 95% CI 2-sided [23.85 to 56.68]
Statistical Analysis 11: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 41.19, 95% CI 2-sided [24.78 to 57.59]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 12]; Test type: Superiority or Other; p = 0.889, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.72, 95% CI 2-sided [-10.89 to 9.45]

13. Secondary Outcome: Duration of Relief
Description: Median participant time for dropping out of the study due to lack of efficacy or receipt of rescue medication, whichever came first.
Time Frame: 0 to 3 hours
Population: Population included all randomized patients that reported a treatment failure or received rescue medication.
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Percentage of participants who withdrew from the study due to lack of efficacy or received rescue medication.
Time Frame: 1, 2, 3 hours post-dose
Population: ITT population included all randomized patients who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
percentage of participants | 0 | 0 | 0

15. Secondary Outcome: Cumulative Percentage of Participants With Complete Relief
Description: Complete relief was defined as a PRR of 4. PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief
Time Frame: 1, 2, & 3 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Number analyzed (Participants) | 91 | 89 | 46
percentage of participants
  1 hour | 0 | 0 | 0
  2 hours | 5.5 | 4.5 | 2.2
  3 hours | 37.4 | 38.2 | 8.7
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.389, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 3.21, 95% CI 2-sided [-3.12 to 9.55]
Statistical Analysis 2: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 8]; Test type: Superiority or Other; p = 0.490, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 2.35, 95% CI 2-sided [-3.69 to 8.39]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; p = 0.764, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 0.98, 95% CI 2-sided [-5.45 to 7.41]
Statistical Analysis 4: Comparison: Ibuprofen Sodium vs Placebo; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 28.71, 95% CI 2-sided [15.72 to 41.70]
Statistical Analysis 5: Comparison: Ibuprofen (Motrin IB) vs Placebo; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 29.37, 95% CI 2-sided [16.19 to 42.56]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 12]; Test type: Superiority or Other; p = 0.898, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.93, 95% CI 2-sided [-15.22 to 13.36]

ADVERSE EVENTS:
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/89 | 0/46
Other Adverse Events (participants affected / at risk) | 0/91 | 0/89 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.